CLINICAL TRIAL: NCT01391988
Title: Prospective Trial Comparing the Use of Conventional Electric Scalpel and Harmonic Scalpel in Mastectomy
Brief Title: Trial Comparing Electric and Harmonic Scalpel in Mastectomy
Acronym: Harmonic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 133/2008 HCB
Record Dates: First submitted 2011-06-24; First posted 2011-07-12 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Complication, Postoperative
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electric Scalpel Mastectomy (Active Comparator): Radical mastectomy with electric scalpel
  Interventions: Procedure: Electric scalpel
- Harmonic scalpel mastectomy (Experimental): Radical Mastectomy with harmonic scalpel
  Interventions: Procedure: Harmonic scalpel

INTERVENTIONS:
Procedure: Electric scalpel — Radical mastectomy with electric scalpel. Electric scalpels were calibrated at 40 watts of cutting and coagulation power.
  Arms: Electric Scalpel Mastectomy
Procedure: Harmonic scalpel — Radical mastectomy with harmonic scalpel. Harmonic GEN04 generator calibrated at power leve 3 and 5, using the HP054 handpiece and HF 105 curved blade
  Arms: Harmonic scalpel mastectomy

SUMMARY:
Prospective trial comparing post-operative complications and seroma formation after mastectomy in patients with breast cancer, using conventional electric scalpel and harmonic scalpel.

DETAILED DESCRIPTION:
The population of this study was formed by women aged older than 18 years old, with breast carcinoma (ductal ou lobular) at any stage, form whom modified radical mastectomy is proposed. Patients were excluded if the present blood dyscrasia, collagen diseases, known uncontrolled chronic disease, infections (mammary or axillary, ulcerated tumors and pregnancy. The women were submitted to modified radical mastectomy consecutive allocated in electric scalpel group and the other group with harmonic scalpel.

Electric scalpels were calibrated at 40 watts of cutting and coagulation power and harmonic scalpel with a GEN04 generator calibrated at power levels 3 and 5, using the HP054 handpiece and HF105 curved blade.

Local postoperative complications analysed were seroma, hematoma, skin necrosis and infection.

ELIGIBILITY:
Women with breast cancer candidate to a radical mastectomy during the year of 2008.

Prospective trial with women stratified consecutive.

Inclusion Criteria:

* Breast carcinoma (ductal or lobular)
* Modified radical mastectomy was the surgery to be realized

Exclusion Criteria:

* Not inclusion criteria
* Blood dyscrasia, collagen diseases, known uncontrolled chronic diseases, infections (mammary or axillary), ulcerated tumors and pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Differences in operative conditions and first week seroma drainage | 1 week.
  Time of the surgery and blood loss volume during surgery. Drain volume postoperative in the first week

SECONDARY OUTCOMES:
Differences in local complication | day 7 and day 14
  Number of participants with adverse events as seroma, hematoma, skin necrosis and infection

CONTACTS AND LOCATIONS:
Overall Officials: Edmundo C Mauad, MD, PhD, Study Director — Director from Barretos Cancer Hospital
Locations (1):
- Hospital de Câncer de Barretos., Barretos, São Paulo, Brazil

REFERENCES:
- [Background] Lumachi F, Brandes AA, Burelli P, Basso SM, Iacobone M, Ermani M. Seroma prevention following axillary dissection in patients with breast cancer by using ultrasound scissors: a prospective clinical study. Eur J Surg Oncol. 2004 Jun;30(5):526-30. doi: 10.1016/j.ejso.2004.03.003. PMID 15135481
- [Background] Lumachi F, Burelli P, Basso SM, Iacobone M, Ermani M. Usefulness of ultrasound scissors in reducing serous drainage after axillary dissection for breast cancer: a prospective randomized clinical study. Am Surg. 2004 Jan;70(1):80-4. PMID 14964555
- [Background] Kozomara D, Galic G, Brekalo Z, Sutalo N, Kvesic A, Soljic M. A randomised two-way comparison of mastectomy performed using harmonic scalpel or monopolar diathermy. Coll Antropol. 2010 Mar;34 Suppl 1:105-12. PMID 20402305
- [Background] Kurtz SB, Frost DB. A comparison of two surgical techniques for performing mastectomy. Eur J Surg Oncol. 1995 Apr;21(2):143-5. doi: 10.1016/s0748-7983(95)90171-x. PMID 7720886
- [Background] Deo SV, Shukla NK, Asthana S, Niranjan B, Srinivas G. A comparative study of modified radical mastectomy using harmonic scalpel and electrocautery. Singapore Med J. 2002 May;43(5):226-8. PMID 12188072
- [Background] Galatius H, Okholm M, Hoffmann J. Mastectomy using ultrasonic dissection: effect on seroma formation. Breast. 2003 Oct;12(5):338-41. doi: 10.1016/s0960-9776(03)00110-3. PMID 14659149
- [Background] Adwani A, Ebbs SR. Ultracision reduces acute blood loss but not seroma formation after mastectomy and axillary dissection: a pilot study. Int J Clin Pract. 2006 May;60(5):562-4. doi: 10.1111/j.1742-1241.2006.00689.x. PMID 16700855
- [Background] Miller E, Paull DE, Morrissey K, Cortese A, Nowak E. Scalpel versus electrocautery in modified radical mastectomy. Am Surg. 1988 May;54(5):284-6. PMID 3364865
- [Derived] Ribeiro GH, Kerr LM, Haikel RL, Peres SV, Matthes AG, Depieri Michelli RA, Bailao A Jr, Fregnani JH, Vieira RA. Modified radical mastectomy: a pilot clinical trial comparing the use of conventional electric scalpel and harmonic scalpel. Int J Surg. 2013;11(6):496-500. doi: 10.1016/j.ijsu.2013.03.013. Epub 2013 Apr 8. PMID 23579255